CLINICAL TRIAL: NCT01085825
Title: The Sensitivity of Manual Versus Electric Vacuum Aspiration to Detect Completed Abortion at Less Than Six Weeks of Pregnancy
Brief Title: Study of the Sensitivity of Manual vs Electric Aspiration to Detect Completed Early Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood of Greater New York (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PPNYC 001
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Induced Abortion
Keywords: induced abortion; termination of pregnancy; manual vacuum aspiration; electric vacuum aspiration
MeSH Terms: interventions — Fumigant 93

ARMS (2):
- Manual Vacuum Aspiration (Active Comparator)
  Interventions: Procedure: D & C abortion
- Electric Vacuum Aspiration (Active Comparator)
  Interventions: Procedure: D & C abortion

INTERVENTIONS:
Procedure: D & C abortion — Participants will be randomized to receive their abortion using either manual vacuum aspiration or electric vacuum aspiration.

SUMMARY:
With sensitive urine pregnancy tests, women are now able to confirm very early pregnancies. However, approximately one third of abortion facilities do not offer abortions at less than six weeks of pregnancy. Providers may be concerned that they will be unable to identify products of conception (POCs) in uterine aspirates after early abortion and about the time, cost and risk associated with following serum hCG levels when completed abortion cannot be confirmed by gross inspection. Many providers believe that manual vacuum aspiration (MVA) causes less destruction of pregnancy tissue and therefore may increase the likelihood of identifying POCs on gross inspection. No published reports specifically compare MVA to electric vacuum aspiration (EVA) for the detection of complete products of conception and none compare MVA and EVA at less than 6 weeks of pregnancy. We, the investigators, propose to conduct a randomized controlled trial comparing the sensitivity of MVA to EVA for the detection of completed abortion in 500 women with pregnancies of less than 6 weeks gestation at a large inner city family planning center. We will measure positive identification of POCs on gross inspection in patients subsequently shown to have completed abortions. We hypothesize that the rate of true positive detection of POCs will be higher in dilation and curettage (D&C) using MVA than EVA.

ELIGIBILITY:
Inclusion Criteria:

* gestational sac size <12 mm or no visible sac (with positive pregnancy test) day of surgical abortion
* no medical contraindications to outpatient abortion at study site

Exclusion Criteria:

* not able to consent
* suspected ectopic pregnancy (pelvic mass, unilateral pain, or detection on ultrasound), suspected molar pregnancy, or no sac and vaginal bleeding suspicious for completed spontaneous abortion
* failed medication abortion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, MPH, Principal Investigator — Planned Parenthood of Greater New York
Locations (1):
- Planned Parenthood of New York City - Margaret Sanger Center, New York, New York, United States

REFERENCES:
- [Derived] Dean G, Colarossi L, Porsch L, Betancourt G, Jacobs A, Paul ME. Manual compared with electric vacuum aspiration for abortion at less than 6 weeks of gestation: a randomized controlled trial. Obstet Gynecol. 2015 May;125(5):1121-1129. doi: 10.1097/AOG.0000000000000787. PMID 25932839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled a total of 500 women from April 22, 2010 to October 14, 2011; 252 women were randomized to MVA and 248 to EVA.
Period: Overall Study
Arm/Group | Manual Vacuum Aspiration | Electric Vacuum Aspiration
Started | 252 (1st participant enrolled) | 248
Completed | 251 | 247
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Vacuum Aspiration | Electric Vacuum Aspiration | Total
Number analyzed (Participants) | 252 | 248 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (5) | 25.4 (5) | 25.4 (5)
Gender [Count of Participants; unit: Participants]
  Female | 252 | 248 | 500
  Male | 0 | 0 | 0
Mean sac diameter [Mean (Standard Deviation); unit: mm] | 8.0 (2.4) | 7.8 (2.3) | 7.9 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Accurate Confirmation of Completed Abortion
Description: Accurate confirmation of completed abortion, as determined by urine pregnancy test at following, appropriately falling serum hCG levels, or patient report of returned menses
Time Frame: 2 weeks - 6 months
Measure: Number; unit: participants
Arm/Group | Manual Vacuum Aspiration | Electric Vacuum Aspiration
Number analyzed (Participants) | 251 | 247
participants | 182 | 164
Statistical Analysis 1: Comparison: Manual Vacuum Aspiration vs Electric Vacuum Aspiration; Test type: Superiority or Other; p = .13, Chi-squared

ADVERSE EVENTS:
Arm/Group | Manual Vacuum Aspiration | Electric Vacuum Aspiration
Serious Adverse Events (participants affected / at risk) | 0/252 | 0/248
Other Adverse Events (participants affected / at risk) | 0/252 | 0/248

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes